CLINICAL TRIAL: NCT02065973
Title: An Open-Label, Phase I, Escalating Dose Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of PDS0101 in Subjects With Cervical Intraepithelial Neoplasia (CIN) and High-risk Human Papillomavirus (HPV) Infection
Brief Title: An Open-Label, Phase I, Escalating Dose Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of PDS0101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PDS Biotechnology Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: U10-02-11-001
Record Dates: First submitted 2014-02-16; First posted 2014-02-19 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: High-risk HPV Infection and Biopsy-proven CIN1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Low Dose) (Active Comparator): The group will receive the lowest dose of the vaccine
  Interventions: Biological: R-enantiomer of 1,2-dioleoyl-3-trimethylammonium-propane chloride + Peptides from HPV-16 E6 and E7
- Cohort 2 (Mid Dose) (Active Comparator): The Group will receive the middle dose of the vaccine
  Interventions: Biological: R-enantiomer of 1,2-dioleoyl-3-trimethylammonium-propane chloride + Peptides from HPV-16 E6 and E7
- Cohort 3 (High Dose) (Active Comparator): The Group will receive the highest dose of vaccine to be tested
  Interventions: Biological: R-enantiomer of 1,2-dioleoyl-3-trimethylammonium-propane chloride + Peptides from HPV-16 E6 and E7

INTERVENTIONS:
Biological: R-enantiomer of 1,2-dioleoyl-3-trimethylammonium-propane chloride + Peptides from HPV-16 E6 and E7

SUMMARY:
Phase I, open-label, sequential-cohort, ascending multiple-dose study to evaluate the safety and tolerability of escalating doses of PDS0101 in female subjects with high-risk HPV infection and biopsy-proven CIN1. The study will include 3 cohorts of 3 to 6 subjects each based on a modified "3 + 3" dose-escalation study design. The study will be initiated with Cohort 1 and progress through Cohort 3, with each subsequent cohort receiving a higher dose of PDS0101. Successive cohorts will receive a constant dose of HPV-16 E6 and E7 peptides. All subjects will receive 3 vaccinations SC given approximately 21 days apart. Dosing and dose escalation will be based on safety evaluation for determination of potential dose-limiting toxicity (DLT).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to initiation of any study-related procedures;
2. Nonlactating female between the ages of 21 to 65 years, inclusive;
3. Non-childbearing potential (defined as surgically sterile or at least 2 years postmenopausal) or practicing effective contraception (defined as 2 concurrent methods of contraception, 1 of which is a barrier method) and agrees to continue using effective contraception throughout the duration of the study;
4. Not pregnant based on a negative result on a serum human chorionic gonadotropin (HCG) test at screening Visit 1 and a negative urine pregnancy test prevaccination at Visit 2 (and at subsequent vaccination visits);
5. Pap test documenting atypical squamous cells of undetermined significance (ASCUS)/HPV+, atypical squamous cells high grade (ASC-H), low-grade squamous intraepithelial lesion (LSIL), or high-grade squamous intraepithelial lesion (HSIL) within 4 months prior to screening Visit 1;
6. History of pathologically confirmed CIN1 by colposcopically-directed punch biopsy, within 12 weeks prior to administration of first study vaccination (CIN 2/3 subjects will not be eligible);
7. For the diagnosis of CIN1, has a documented satisfactory colposcopy, ie, the entire lesion as well as the entire squamocolumnar junction is visualizible by colposcopy;
8. Confirmed high-risk HPV infection by a commercially available high-risk DNA assay (eg, Hybrid Capture II [Qiagen]);
9. Good health with adequate hematologic, renal, hepatic, and cardiac function, as determined by the Investigator, based upon medical history, physical examination, and laboratory test results at the screening visit (Visit 1):

   * Bone marrow function: absolute neutrophil count ≥1,500/µL, and platelets ≥ 100,000/ µL;
   * Renal function: creatinine ≤ 1.5 x institutional upper limit of normal (ULN);
   * Hepatic function: total bilirubin ≤ 1.5 x ULN (Common Terminology Criteria for AEs [CTCAE] v4.0 grade 1) except patients with Gilbert's disease (up to 5.0 mg/dL). Aspartate aminotransferase (AST) and alkaline phosphatase ≤ 2.5 x ULN.
   * Normal Cardiac function: as assessed by history and physical exam.

Exclusion Criteria:

1. Atypical endometrial or glandular cells or evidence of invasive cervical carcinoma on cervical biopsy;
2. Previous history of cancer, other than adequately treated basal cell or Stage 1 squamous cell carcinoma of the skin;
3. Current recognized immunodeficiency disease, including infection with HIV, cellular immunodeficiencies, hypogammaglobulinemia, or dysgammaglobulinemia, or hereditary or congenital immunodeficiencies.
4. Received immunotherapy (eg, IFNs, tumor necrosis factor, interleukins, or biological response modifiers [granulocyte-macrophage colony-stimulating factor, granulocyte colony-stimulating factor, macrophage colony-stimulating factor]) within 30 days prior to administration of the first study vaccination;
5. Serious, concomitant disorder, including active systemic infection requiring treatment, in the opinion of the investigator;
6. Currently receiving or has received treatment with systemic steroids in the following dosages within 30 days prior to administration of the first study vaccination.

   * Chronic or long-term corticosteroids: ≥0.5 mg/kg/day of oral prednisolone or equivalent
   * Sporadic corticosteroids: ≥1 mg/kg/day of oral prednisolone or equivalent for 2 or more short courses of > 3 days
   * Note: Current or recent use of intra-articular, topical or inhaled glucocorticoid therapy is acceptable;
7. Other condition or prior therapy that, in the opinion of the Investigator, compromises the subject's welfare or may confound study results;
8. Participation in another investigational study concurrently or use of another investigational drug within 6 months prior to administration of the first study vaccination;
9. Previously enrolled in this study.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluation or determination of adverse events following vaccination | Days 1-133

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Suffolk Obstetrics & Gynecology, Port Jefferson, New York
  - Montefiore Medical Center, The Bronx, New York